CLINICAL TRIAL: NCT05808244
Title: A Randomised Controlled Study on Feasibility of Tele-group Cognitive Behavioural Family Intervention (tgCBFI) for People With Schizophrenia and Their Families
Brief Title: Tele-group Cognitive Behavioural Family Intervention (tgCBFI) for People With Schizophrenia and Their Families
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other); Queen Mary Hospital, Hong Kong (Other); Kowloon Hospital, Hong Kong (Other); Nethersole Institute of Continuing Holistic Health Education (Unknown)
Responsible Party: Principal Investigator, Dennis Chak Fai Ma, Clinical Associate (Mental Health), The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tgCBFI
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tgCBFI (Experimental)
  Interventions: Behavioral: tgCBFI; Behavioral: Usual psychiatric care
- Usual psychiatric care (Active Comparator)
  Interventions: Behavioral: Usual psychiatric care

INTERVENTIONS:
Behavioral: tgCBFI — Six weekly sessions CBT-based family intervention programme
  Arms: tgCBFI
Behavioral: Usual psychiatric care — Integrated community psychiatric care with medical follow-up

SUMMARY:
This mixed-method study aims to examine the feasibility of delivering tgCBFI programme to dyads of people with schizophrenia and their family caregivers, and generate preliminary evidence on the effectiveness of tgCBFI in reducing expressed emotion. The research questions are as follows.

1. What are the feasibility, acceptability, and safety of conducting a tele-group CBFI programme for people with schizophrenia and their family caregivers?
2. What effect does tgCBFI have on the expressed emotion experienced by adults with schizophrenia and the caregiving experience of their family caregivers at posttreatment and 12-week after completion of the programme?
3. What effect does tgCBFI have on the positive and negative symptoms of adults with schizophrenia and the perceived care burden and level of mood disturbance of their family caregivers at posttreatment, and 12-week after completion of the programme?

ELIGIBILITY:
Inclusion Criteria:

Service users

* diagnosis of schizophrenia-spectrum disorders, based on ICD-10 made by the treating clinicians
* aged 18 to 64
* able to communicate in Cantonese

Family caregivers

* aged 18 or above
* able to communicate in Cantonese
* live with service users

Exclusion Criteria:

Service users

* have co-morbidity of learning disability, organic/neurological conditions, or substance misuse disorder
* live in hostel

Family caregivers

-have active psychiatric conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Level of service satisfaction of service users and family caregivers | Immediate posttreatment
Feasibility, acceptability, and safety of the programme | Throughout the whole programme

SECONDARY OUTCOMES:
Perceived expressed emotion of service users | up to 12-week follow up
Positive and negative symptoms of service users | up to 12-week follow up
Mood disturbance of family caregivers | up to 12-week follow up
Perceived care burden of family caregivers | up to 12-week follow up
Qualitative feedback from service users and family caregivers | Immediate posttreatment